CLINICAL TRIAL: NCT04219566
Title: Pilot Study to Demonstration of Safety and Efficacy of VeSTAL Sleep Device in Human Subjects: Randomized Study of VeSTAL Compared to Sham Control as a Means of Improving Sleep as Determined by ISI Scores
Brief Title: Vestibular Nerve Stimulation to Improve Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: RD Gardi Medical College (Unknown); Compliance Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVS001S
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Insomnia; Sleep; Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Nursing staff, Co-coordinators, Outcomes Assessor and any other study staff who have contact with the subject)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active VeNS (Active Comparator): The VeSTAL device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day in the period immediately prior to sleep onset.
  Interventions: Device: VeNS
- Sham VeNS (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. However, it does not deliver vestibular stimulation to users. device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day in the period immediately prior to sleep onset.
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: VeNS — Non-invasive electrical vestibular nerve stimulation
  Arms: Active VeNS
Device: Placebo device — Sham non-invasive electrical vestibular nerve stimulation
  Arms: Sham VeNS

SUMMARY:
A randomized, double blind sham controlled clinical trial to evaluate the efficacy of vestibular nerve stimulation (VeNS) compared to a sham control a as a means of improving sleep as measured by ISI scores and EEG recordings

The purpose of this investigation device study is to collect data that will be used to design appropriate pivotal studies that can be used for regulatory submissions, primarily in the United States of America (USA), but it may also be used to support submissions in other regions, including the European Union (EU).

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Both genders
* Ages 18-24 years inclusive
* Score above 14 in the insomnia severity index questionnaire
* Willingness to participate in the study.

Exclusion Criteria:

* Use sleep medication
* Ear problems
* Under any kind of treatment
* Practicing sleep improving techniques
* Any other significant health-related problems.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) Scores | Day 0, Day 7, Day 14, Day 21, Day 28
  ISI scores will be measured during the study and will be compared to baseline readings taken prior to intervention. Insomnia Severity Index scores range from 0 to 28. Scores greater than 15 indicate clinical insomnia.

SECONDARY OUTCOMES:
EEG Assessment | Day 0, Day 28
  EEG power in alpha band
Depression Anxiety Stress Scales (DASS) Assessment | Day 0, Day 7, Day 14, Day 21, Day 28
  DASS will be measured during the study and will be compared to baseline readings taken prior to intervention. DASS is scored from 0 to 42 with higher scores indicating more symptoms.
WHO Quality of Life (WHOQOL) Assessment | Day 0, Day 7, Day 14, Day 21, Day 28
  QOL will be measured during the study and will be compared to baseline readings taken prior to intervention. WHOQOL is scored from 0 to 100 with higher scores indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Sailesh, Principal Investigator — RD Gardi Medical College
Locations (1):
- RD Gardi Medical College, Ujjain, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Data will be transferred in an encrypted PDF format. Trial staff will be given direction on how to share the trial data and given access to one specific section of a controlled cloud service which is controlled via role based access. Once they have authenticated with the service and the service verifies that they have the correct role to access the system they will be directed to a single webpage within the application where they will be able to upload the encrypted PDF. This PDF is generated on the fly and is therefore not stored in another location that could become compromised. Generating the PDF on the fly means that the source data is extracted from the database, processed and delivered in the context of a single request. These data will be transferred for each subject when they complete participation in the study.